CLINICAL TRIAL: NCT07396090
Title: A Clinical Study of Safety, Immunogenicity and Preliminary Efficacy of mKRAS Antigen-Loaded eDCs (CAT-101) Monotherapy or Plus Tislelizumab (Anti-PD-1 mAb) in KRAS-G12C/D/R/V-Mutated Advanced Pancreatic Cancer and Other Solid Tumors
Brief Title: Study of KRAS-Specific Vaccine in Patients With KRAS-Mutated Solid Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, NING_LI, Chief, Office of Clinical Trial Center, CancerIHCAMS, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAT-101
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group (Experimental): mKRAS antigen-loaded engineered dendritic cells (eDCs, designated as CAT-101)
  Interventions: Biological: eDC-KRAS vaccine; Drug: Tislelizumab

INTERVENTIONS:
Biological: eDC-KRAS vaccine — intravenous injection
Drug: Tislelizumab — intravenous injection

SUMMARY:
The purpose of this study is to evaluate the safety, immunogenicity and preliminary efficacy of engineered dendritic cells（eDCs）loaded with mKRAS antigen (CAT-101) alone or in combination with Tislelizumab (anti-PD-1 monoclonal antibody) among participants with KRAS-G12C/D/R/V mutated advanced pancreatic cancer and other solid tumors.

DETAILED DESCRIPTION:
The primary objective of this study is to systematically evaluate the safety profile, immunogenicity, and preliminary clinical efficacy of mKRAS antigen-loaded engineered dendritic cells (eDCs, designated as CAT-101), administered either as monotherapy or in combination with Tislelizumab (an anti-PD-1 monoclonal antibody), in patients with KRAS-G12C/D/R/V-mutated advanced pancreatic cancer and other refractory solid tumors. Secondary objectives include exploring the correlation between treatment-induced immune responses and clinical outcomes, as well as characterizing the optimal administration regimen for this combination therapy.

ELIGIBILITY:
Inclusion Criteria:（1）Age 18-75 years，Male or female ； （2）Participants with ECOG score of 0-1 and the life expectancy ≥6 months； （3）Sufficient organ function as defined by the following criteria: creatinine clearance of ≥45 mL/min;Serum AST and serum ALT, ≤3.0 x ULN (≤5 x ULN for patients with liver metastases); Total bilirubin (TBIL) and alkaline phosphatase (AKP or ALP) ≤2.0 × ULN (except for congenital hyperbilirubinemia, such as Gilbert syndrome, the direct bilirubin may be ≤1.5 × ULN); for patients with liver and/or bone metastases, alkaline phosphatase ≤5.0 × ULN; Left ventricular ejection fraction ≥45% (by echocardiography or MUGA) (4) pregnancy test for women must be negative, and or must not be breastfeeding; participants with childbearing potential must agree to use effective contraception from the signing of the informed consent form until 1 year after the use of the study drug; (5) Willing to sign the informed consent form (ICF); （6）HLA-A*1101+ Participants with histologically confirmed advanced solid tumors (such as pancreatic ductal adenocarcinoma, non-small cell lung cancer, etc.) and harboring at least one of the targeted KRAS mutants （G12C/D/R/V）; (7)Participants who have failed standard treatment or who have no standard treatment options or who have minimal residual disease (MRD) after standard treatment , as well as those have unresectable locally advanced or metastatic solid tumors but currently unsuitable for standard treatment.

(8) Participants must have measurable lesions detected by computed tomography (CT) or magnetic resonance imaging (MRI) (according to iRECIST criteria);

-

Exclusion Criteria:(1) Patients received other investigational therapy or any chemotherapy, hormonal therapy, targeted therapy, epigenetic therapy, or treatment with invasive investigational medical devices within 4 weeks or 5 half-lives prior to the first vaccination (whichever is shorter):

(2)Patients received proteasome inhibitors and immunomodulators, radiotherapy, or approved Chinese traditional medicine within 2 weeks or 5 half-lives prior to the first vaccination(whichever is shorter), (3) patients with meningeal, brainstem, or spinal cord metastases and/or compression, or active central nervous system (CNS) metastases; Participants with asymptomatic brain metastases within 4 weeks before the first vaccination and who do not require steroid treatment for at least 14 days are eligible for enrolment.

(4) patients with active second primary malignancy; however, patients received curative treatment and without known active disease for ≥2 years or non-melanoma skin cancer patients who received adequately treatment and with no evidence of disease will be eligible for study entry (5) patients with severe uncontrolled infection (bacterial, viral, fungal, etc.) during the screening period; (6) known positive test results for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood hepatitis B virus (HBV) DNA titer above the normal range or positive for hepatitis C virus (HCV) antibody with peripheral blood HCV RNA titer above the normal range or positive for human immunodeficiency virus (HIV) antibody; positive syphilis test within 6 months prior to the vaccinations.

(7)Patients with symptomatic heart failure or other cardiac diseases such as severe arrhythmias:

* New York Heart Association (NYHA) Class III or IV congestive heart failure;
* Myocardial infarction or coronary artery bypass graft (CABG) or coronary stent implantation within ≤6 months prior to signing the ICF;
* Clinically significant ventricular arrhythmia, or history of unexplained syncope (excluding vasovagal or dehydration-related causes);
* History of severe non-ischemic cardiomyopathy; （8）patients with other diseases, including:
* Primary immunodeficiency;
* Stroke or seizure within 6 months prior to screening;
* Significant clinical evidence of dementia or altered mental status;
* Parkinson's disease or Parkinson-like movement disorders or history thereof;
* Uncontrolled hypothyroidism or hyperthyroidism; (9)Surgery within 2 weeks prior to the vaccination or planned surgery within 2 weeks after the vaccination, excluding local anesthesia; （10）Uncontrolled hypertension, hypercalcemia, or diabetes; （11）Vaccination with live attenuated vaccines within 1 month prior to the first infusion; （12） Patients who have undergone long-term systemic corticosteroid therapy; （13）Known severe allergic reactions to eDC products or their formulation components (e.g., albumin, IL-2) （14）eDC-KRAS preparation failed; （15）Researchers believe that other reasons are not suitable for clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to 24 months
  Adverse events defined as the number of participants with adverse events according to CTCAE v5.0.

SECONDARY OUTCOMES:
Objective Response Rate | up to 24 months
  The proportion of patients achieving a predefined reduction in tumor burden as assessed by Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Responses are categorized as complete response (CR, disappearance of all target lesions) or partial response (PR, ≥30% reduction in the sum of target lesion diameters), with ORR calculated as the percentage of patients with CR or PR relative to the total evaluable cohort.
Immunogenicity of eDC-KRAS vaccine | up to 24 months
  Measure vaccine-induced immune response (e.g., antigen-specific T-cell/cytokine responses /lymphocyte subsets changes).
Rate of MRD Clearance | up to 24 months
  The percentage of patients who achieve minimal residual disease (MRD) negativity following treatment, defined as the absence of detectable tumor-specific biomarkers (e.g., circulating tumor DNA, tumor-associated antigens) or malignant cells in peripheral blood, bone marrow, or other relevant biological samples, using a validated, high-sensitivity detection assay.
Disease Control Rate (DCR) | up to 24 months
  The percentage of patients whose disease is controlled, encompassing those with complete response (CR), partial response (PR), and stable disease (SD, no significant increase or decrease in target lesion size per RECIST v1.1 criteria) for a minimum of the predefined evaluation period. DCR reflects the treatment's ability to inhibit tumor progression in the evaluable patient population.
Duration of Relief | up to 24 months
  The time interval from the first documentation of a clinically meaningful reduction in cancer-related symptoms (e.g., pain, fatigue, dyspnea) to the recurrence of symptoms or initiation of subsequent anti-tumor therapy. Symptom assessment is based on validated patient-reported outcome (PRO) scales or clinician-administered symptom rating tools, with relief defined by a predefined threshold of symptom improvement.
Progress-Free Survival (PFS) | up to 24 months
  The time from treatment initiation to the first documentation of tumor progression (per RECIST v1.1) or death from any cause, whichever occurs first. PFS is measured using standardized imaging assessments performed at predefined time points and is a key endpoint reflecting the treatment's ability to delay disease progression.
Overall Survival (OS) | up to 24 months
  The time from treatment initiation to death from any cause. OS is a definitive endpoint that evaluates the treatment's impact on patient survival, with follow-up conducted until patient death or the end of the study's observation period.
Tumor Markers Changes | up to 24 months
  The dynamic alterations in the levels of tumor-associated serological or tissue biomarkers (e.g., CA 19-9, CEA, CA 125) measured at baseline and at predefined post-treatment time points. Changes are quantified as the percentage reduction or increase from baseline, with a predefined threshold (e.g., ≥50% reduction) used to define a clinically significant change. These data are analyzed to explore correlations with clinical response and disease progression.